CLINICAL TRIAL: NCT07092215
Title: Mechanisms of Pain Hypersensitivity in a Human Skin Inflammation Model - A Double-blind, Randomized, Placebo-controlled Crossover Study
Brief Title: Mechanisms of Pain Hypersensitivity in a Human Skin Inflammation Model
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stefan Heber (Other)
Responsible Party: Sponsor-Investigator, Stefan Heber, Principal Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EK1692/2024
Record Dates: First submitted 2025-06-11; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pain
Keywords: Inflammation; Skin; Pain model; Hyperalgesia; RAGE; Azeliragon; TLR4; Resatorvid; TRPV1; BCTC
MeSH Terms: conditions — Pain; Inflammation; Hyperalgesia | interventions — Lipopolysaccharides; azeliragon; ethyl 6-(N-(2-chloro-4-fluorophenyl)sulfamoyl)cyclohex-1-ene-1-carboxylate

STUDY DESIGN:
Intervention Model Description: The study is designed as a double-blind, randomized, placebo-controlled crossover study. The study design involves 10 groups. The low local dose, which does not spread to other test sites as well as the short duration of biological effects induced by pain, excludes biological carry over effects. To prevent bias from psychological carryover effects, multiples of 10 participants are tested using a Latin squares balanced design according to Williams (https://adsabs.harvard.edu/full/1949ausra...2..149w). For each participant, one of 10 pre- specified sequences is randomly selected and removed from the pool.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To ensure double-blind conditions, all solutions are prepared and numbered by an independent laboratory technician who is not involved in the experiment. Both the participants and the experimenter are blinded to the injected substances (LPS, Azeliragon, Resatorvid, BCTC) and to whether solutions contain neutral or acidic solutions for the acid-induced pain model. Familiarization injections are administered unblinded for safety and tolerability assessment. Blinding is maintained until the end of each subject's participation. Randomization sequences are generated and stored separately and are only accessible to unblinded personnel in case of emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Sequence #01 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. SIF (neutral pH)
  2. SIF (acidic pH)
  3. LPS + RES (acidic pH)
  4. SIF (acidic pH + BCTC)
  5. LPS + RES (neutral pH)
  6. LPS (neutral pH)
  7. LPS + AZE (acidic pH)
  8. LPS (acidic pH)
  9. LPS + AZE (neutral pH) 10. LPS (acidic pH + BCTC)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #03 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. SIF (acidic pH + BCTC)
  2. LPS (neutral pH)
  3. SIF (acidic pH)
  4. LPS (acidic pH)
  5. SIF (neutral pH)
  6. LPS (acidic pH + BCTC)
  7. LPS + RES (acidic pH)
  8. LPS + AZE (neutral pH)
  9. LPS + RES (neutral pH) 10. LPS + AZE (acidic pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #04 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. LPS (neutral pH)
  2. LPS (acidic pH)
  3. SIF (acidic pH + BCTC)
  4. LPS (acidic pH + BCTC)
  5. SIF (acidic pH)
  6. LPS + AZE (neutral pH)
  7. SIF (neutral pH)
  8. LPS + AZE (acidic pH)
  9. LPS + RES (acidic pH) 10. LPS + RES (neutral pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #05 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. LPS (acidic pH)
  2. LPS (acidic pH + BCTC)
  3. LPS (neutral pH)
  4. LPS + AZE (neutral pH)
  5. SIF (acidic pH + BCTC)
  6. LPS + AZE (acidic pH)
  7. SIF (acidic pH)
  8. LPS + RES (neutral pH)
  9. SIF (neutral pH) 10. LPS + RES (acidic pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #06 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. LPS (acidic pH + BCTC)
  2. LPS + AZE (neutral pH)
  3. LPS (acidic pH)
  4. LPS + AZE (acidic pH)
  5. LPS (neutral pH)
  6. LPS + RES (neutral pH)
  7. SIF (acidic pH + BCTC)
  8. LPS + RES (acidic pH)
  9. SIF (acidic pH) 10. SIF (neutral pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #07 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. LPS + AZE (neutral pH)
  2. LPS + AZE (acidic pH)
  3. LPS (acidic pH + BCTC)
  4. LPS + RES (neutral pH)
  5. LPS (acidic pH)
  6. LPS + RES (acidic pH)
  7. LPS (neutral pH)
  8. SIF (neutral pH)
  9. SIF (acidic pH + BCTC) 10. SIF (acidic pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #08 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. LPS + AZE (acidic pH)
  2. LPS + RES (neutral pH)
  3. LPS + AZE (neutral pH)
  4. LPS + RES (acidic pH)
  5. LPS (acidic pH + BCTC)
  6. SIF (neutral pH)
  7. LPS (acidic pH)
  8. SIF (acidic pH)
  9. LPS (neutral pH) 10. SIF (acidic pH + BCTC)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #09 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. LPS + RES (neutral pH)
  2. LPS + RES (acidic pH)
  3. LPS + AZE (acidic pH)
  4. SIF (neutral pH)
  5. LPS + AZE (neutral pH)
  6. SIF (acidic pH)
  7. LPS (acidic pH + BCTC)
  8. SIF (acidic pH + BCTC)
  9. LPS (acidic pH) 10. LPS (neutral pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #10 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. LPS + RES (acidic pH)
  2. SIF (neutral pH)
  3. LPS + RES (neutral pH)
  4. SIF (acidic pH)
  5. LPS + AZE (acidic pH)
  6. SIF (acidic pH + BCTC)
  7. LPS + AZE (neutral pH)
  8. LPS (neutral pH)
  9. LPS (acidic pH + BCTC) 10. LPS (acidic pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH
- Sequence #02 (Experimental): Participants receive 10 intradermal injetions at time point -4.5h, of which 3 contain no substance (SIF), 3 contain LPS, 2 contain LPS + AZE and 2 contain LPS + RES. This is followed by laser speckle imaging (all skin spots), mechanical stimulation (all skin spots) and injection of neutral OR acidic solutions, containing OR not containing BCTC (stated in parantheses) at time point 0. The order is as follows:
  1. SIF (acidic pH)
  2. SIF (acidic pH + BCTC)
  3. SIF (neutral pH)
  4. LPS (neutral pH)
  5. LPS + RES (acidic pH)
  6. LPS (acidic pH)
  7. LPS + RES (neutral pH)
  8. LPS (acidic pH + BCTC)
  9. LPS + AZE (acidic pH) 10. LPS + AZE (neutral pH)
  Interventions: Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH; Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng / SIF neutral pH; Drug: LPS 5 ng / SIF acidic pH; Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM; Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH; Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH; Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH

INTERVENTIONS:
Drug: Synthetic interstitial fluid (SIF) / SIF neutral pH — Intradermal injection of SIF at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with neutral pH (pH 7.4)
Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH — Intradermal injection of SIF at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with acidic pH (pH 7.4 to pH 5.7)
Drug: Synthetic interstitial fluid (SIF) / SIF acidic pH + BCTC 1 µM — Intradermal injection of SIF at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with acidic pH (pH 7.4 to pH 5.7), containing BCTC 1 µM
Drug: LPS 5 ng / SIF neutral pH — Intradermal injection of LPS 5 ng at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with neutral pH (pH 7.4)
Drug: LPS 5 ng / SIF acidic pH — Intradermal injection of LPS 5 ng at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with acidic pH (pH 7.4 to pH 5.7)
Drug: LPS 5 ng / SIF acidic pH + BCTC 1 µM — Intradermal injection of LPS 5 ng at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with acidic pH (pH 7.4 to pH 5.7), containing BCTC 1 µM
Drug: LPS 5 ng + Azeliragon 100 µM / SIF neutral pH — Intradermal injection of LPS 5 ng + Azeliragon 100 µM at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with neutral pH (pH 7.4)
Drug: LPS 5 ng + Azeliragon 100 µM / SIF acidic pH — Intradermal injection of LPS 5 ng + Azeliragon 100 µM at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with acidic pH (pH 7.4 to 5.7)
Drug: LPS 5 ng + Resatorvid 10 µM / SIF neutral pH — Intradermal injection of LPS 5 ng + Resatorvid 10 µM at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with neutral pH (pH 7.4)
Drug: LPS 5 ng + Resatorvid 10 µM / SIF acidic pH — Intradermal injection of LPS 5 ng + Resatorvid 10 µM at time point -4.5h, followed by laser speckle imaging, mechanical stimulation and intradermal injection of SIF with neutral pH (pH 7.4 to pH 5.7)

SUMMARY:
The main goal of this double-blind, randomized, placebo-controlled crossover study is to understand the molecular mechanisms of inflammation-induced increased pain sensitivity (hyperalgesia). These mechanisms are studied using a recently established human model of skin inflammation that mimics aspects of skin infection. A localized inflammatory response in the skin of healthy volunteers is elicited by locally injecting a small, safe dose of Lipopolysaccharide (LPS), a major component of gram-negative bacteria.

The study addresses three key research questions:

* Role of RAGE: To investigate if certain inflammatory effects of LPS, which contribute to hyperalgesia, are mediated by a signaling pathway involving the RAGE receptor.
* Pain Sensitization: To examine how skin inflammation affects pain caused by acidic stimuli, and to differentiate this from purely mechanical pain.
* Role of TRPV1: To determine if the contribution of the TRPV1 ion channel to acid-induced pain is different in inflamed skin.

Participants will undergo an experimental session 4.5 hours after LPS injection to measure skin blood flow (using laser speckle imaging), mechanical pain sensitivity (using specialized tweezers), and pain induced by injecting a solution, of which the pH is gradually decreasing (acid-induced pain).

The study has minimal risks due to the small, safe doses of substances used ('microdosing') and aims to lay the groundwork for developing new treatments for inflammatory pain conditions.

DETAILED DESCRIPTION:
Inflammation is recognized as a major contributor to both acute and chronic pain conditions. To develop new treatments for inflammatory pain, it is essential to understand the underlying molecular mechanisms. The skin is particularly suitable for such studies due to its accessibility. This study builds on a previously established human skin model that reflects the proinflammatory aspects of skin infection, aiming to investigate the mechanisms of inflammation-induced hyperalgesia, using various painful stimuli.

Skin and soft tissue infections encompass a range of conditions caused by gram-positive and gram-negative bacteria, often involving multiple pathogens. These infections can range from superficial and relatively harmless, like furuncles, to severe and life-threatening, such as necrotizing fasciitis. Lipopolysaccharide (LPS), an immunogen component of gram-negative bacterial cell walls, is commonly used in clinical research. LPS induces a strong immune response and has been safely applied in human studies both intravenously and intradermally. When injected intradermally at doses of 5-15 ng, LPS produces localized inflammatory lesions that resolve within 48 hours and do not cause systemic symptoms (CITs).

LPS acts mainly through Toll-like receptor 4 (TLR4) on immune cells, but also potentially through the receptor for advanced glycation end products (RAGE; CIT), which may directly sensitize sensory neurons (CIT). This study uses co-injection of the RAGE antagonist Azeliragon to explore the role of RAGE in LPS-induced hyperalgesia. The TLR4 antagonist Resatorvid will also be tested by co-injection. Determining the involvement of these signalling pathways could guide the development of future therapeutic agents.

A prior exploratory pilot study (n = 12) mapped the time course and degree of pain hypersensitivity following LPS application using laser speckle imaging to measure hyperemia, a contact heat stimulus to study potential thermal hyperalgesia, tweezers to study potential mechanical hyperalgesia and intradermal acidic injections to study acid-induced pain. The current study builds on this to assess whether LPS-induced hyperalgesia is mediated, at least in part, through RAGE-dependent pathways. In addition, the involvement of transient receptor potential cation channel subfamily V member 1 (TRPV1) in acid-induced pain will be investigated in the inflammation model, by co-injecting TRPV1 antagonist BCTC with the acidified solution. Previous research showed that injection of acidic fluid induces pain in non-inflamed skin, which is fully TRPV1-dependent (CIT), but it remains unclear whether this also applies to an inflamed condition.

Study objective and hypotheses The aim of this study is to elucidate the mechanisms of LPS-induced hyperalgesia, which leads to three independent research questions.

Research Question 1 (Main Research Question): The Role of RAGE in LPS-induced inflammation The mediation of immunogenic effects of LPS via TLR4 has long been established. The question remains whether parts of the proinflammatory effects of LPS are also mediated through an alternative RAGE-dependent signaling pathway, contributing to hyperalgesia. Antagonizing TLR4 serves as a reference. Blood flow provides an objective readout.

Primary Hypothesis: The degree of hyperemia is different in LPS-injected skin spots (3x) compared to LPS-injected skin spots where Azeliragon is co-injected (2x).

Secondary Hypothesis 1: Acid-induced pain is different in LPS-injected skin spots (1x) compared to LPS-injected skin spots where Azeliragon is co-injected (1x).

Secondary Hypothesis 2: Mechanically induced pain is different in LPS-injected skin spots (3x) compared to LPS-injected skin spots where Azeliragon is co-injected (2x).

In the respective comparison groups, the contribution of TLR4 is measured with the antagonist Resatorvid as a reference.

Research Question 2 (Exploratory): Sensitization in the LPS inflammation model This question concerns the pain induced by the injection of increasingly acidic (pH = 7.4 to 5.7) or neutral (pH = 7.4) solutions, differentiating between purely mechanical hyperalgesia and additional hyperalgesia due to acidosis.

The pilot study demonstrated that acid-induced pain in the skin after LPS injection is greater than after control injection. It also showed that mechanically induced pain on the skin after LPS injection is greater than after control injection. However, it remains unclear whether the difference between mechanically and acid-induced pain changes after LPS injection.

Hypothesis (Exploratory): The pain induced by acidosis in addition to mechanically induced pain (by injection into the skin) is greater after LPS injection than after control injection

. Research Question 3 (Exploratory): The Role of TRPV1 in acid-induced pain in the LPS inflammation model The question is whether the proportion of acid-induced pain attributable to TRPV1 activation is altered by LPS-induced inflammation.

Hypothesis (Exploratory): The inhibition of acid-induced pain by adding BCTC to the injection solution is greater after LPS injection than after control injection.

Study design This study is intended for non-therapeutic biomedical research on humans (basic research). It is designed as a double-blind, randomized, placebo-controlled crossover study. The study is performed at the Division of Special Anesthesia and Pain Medicine, AKH Vienna, Vienna, Austria.

Methodology and experimental procedures First, for female participants, pregnancy is excluded by a pregnancy test. In case of a positive test, the participant is excluded and will be compensated for travelling. Before induction of skin inflammation by LPS injection, subjects will be familiarized with the subsequent pain stimuli (mechanical and acid) at two distinct native skin spots. The procedures are fully identical to the test stimulation for mechanical pain and acid-induced pain. The only difference is that it serves only for the subject to get to know the procedure. These stimulations will not be considered in the analysis. Thereafter, LPS ± substances are injected. After a period of 4.5 h, noxious stimuli as in the pilot study are applied. The procedure for determining mechanical hyperalgesia and acid-induced pain remains unchanged; two of the injection solutions will additionally contain BCTC.

Time point 1: Induction of skin inflammation resembling bacterial infection To trigger an inflammatory response resembling infection with gram-negative bacteria in the skin of human subjects, 5 ng of LPS dissolved in 50 µl of SIF, will be injected superficially into premarked skin spots of the volar forearm 4.5h before the application of noxious stimuli using a 30G syringe. The dose of 5 ng of LPS is based on literature (CIT), which was validated in pilot experiments. Each participant receives 10 injections, with 3 control injections and 7 injections containing LPS. In two LPS injections, the RAGE antagonist Azeliragon (100µM) is added, and in another two the TLR4 antagonist Resatorvid (10µM).

Time point 2: Quantification of skin perfusion The degree of hyperemia is quantified by using laser speckle imaging. It can be assumed that the inflamed skin area itself does not systematically vary between spots and subjects. In contrast to that, the distance at which the images are taken may vary between subjects. Therefore, a circular adhesive sticker of a diameter of 2 cm is placed in the center of both forearms as a reference. The subject is then asked not to move the forearm for a few seconds to acquire blood flow and a color image. The same procedure is repeated on the contralateral forearm.

Time point 2: Model of mechanical hyperalgesia Mechanical stimulation of the skin is realized by the use of self-closing cross-over tweezers. The tweezers are customized to have an maximal opening diameter of 6 mm, which fits the total area of erythema arising from the inflammation model used. For stimulation, the levers are opened by squeezing, gently put onto the test site, and closed by releasing. The self-closing property of the tweezers allows applying a standardized pinch to the skin, intensity of the perceived pain is rated by the subject thereafter. All pain ratings are provided on a scale 0-100, where 0 indicates not pain and 100 the maximal imaginable pain. The subjects are positioned and instructed not to look at the test site. For each spot the mechanical sensitivity is tested three times.

Time point 2: Model of acid-induced pain To expose human subjects to a defined nonhazardous intradermal acidic stimulus, the protocols of our two recent studies (continuous injection of constant pHs of 7.0, 6.5, 6.0 or 4.3, respectively) have been further developed to provide a linear decrease from a pH of 7.4 to a pH of 5.7. This is realized by two syringes connected via perfusor lines to a 3-way stopcock, where the solutions are being mixed before intradermal injection through a 30G cannula. The syringes contain SIF with a pH of 7.4 and 5.0, respectively. Over a period of 110 seconds, two programmable pumps stepwise adapt their infusion rates to generate a linear decrease from a pH of 7.4 to a pH of 5.7. The summarized total infusion rate is fixed at 30 ml/h throughout the protocol, which results in a total volume of 0.92 ml administered per injection. As in previous studies, pain is rated every five seconds on a numerical pain rating scale ranging from 0 to 100, whereas 0 represents no pain and 100 the maximum imaginable pain. Stimulation will alternatingly use both forearms. First, the cannula is intradermally inserted into the respective spot (inflamed or non-inflamed) on the volar forearm of the subject and further fixed with Leukoplast to prevent slipping of the stopcock. The infusion and the stopwatch are started simultaneously when no pain (= 0) is reported after cannula insertion. Pain is rated every five seconds until the subject reports no pain for a period of 30 consecutive seconds. A non-acidic stimulus is obtained by filling both syringes with solutions of a pH of 7.4.

Applied substances, dosage and administration Synthetic interstitial fluid (SIF) To closely mimic extracellular fluid, we previously used a synthetic interstitial fluid (SIF) (CIT). To reach a physiological buffer capacity, histidine (pKa=6.0) is added at 22.0 mM. This SIF variant allows for a stable pH in the range of 5.0 to 7.4 and contains the following (in mmol/l): NaCl 113.8, KCl 3.5, Na2HPO4 1.7, MgSO2×7H2O 0.7, sodium gluconate 9.6, glucose 5.0, sucrose 7.6, CaCl2×2H2O 1.5, Histidine 22.0. The calculated osmolarity is 300 mosmol/l. All fluids injected are diluted in SIF adjusted to a pH of 7.4. For the acid induced pain model, SIF is adjusted to a pH of 7.4 and 5.0, respectively.

Lipopolysaccharide (LPS) Lipopolysaccharide (LPS; Molecular formula: C205H366N3O117P5; 4900 g/mol) is a major constituent of the cell wall of gram-negative bacteria. It is acquired from List Biological Laboratories as a highly purified molecule obtained from Escherichia coli O113, which has been shown to be safe in humans (CIT). Notably, List Biological Laboratories was commissioned by the NIH to manufacture GMP grade reference endotoxin (CIT). According to the corresponding author, the same source has been used for two of the above mentioned studies on intradermal LPS challenge (CITs). In this study, applying a dose of 5 ng per injection, 7 injections of LPS will result in a total dose of 35 ng, which is in the range of total doses used in previous intradermal trials and far below the total doses injected in intravenous trials (up to 300 ng). None of our preliminary experiments with repeated injections of LPS have indicated systemic adverse effects.

Resatorvid This TLR4 antagonist is co-injected with LPS at a dose of 2 x 0.18 µg = 0.36 µg. Resatorvid has undergone Phase III trials (daily doses of 1.2 or 2.4 mg/kg intravenously for 4 days, equivalent to daily doses of 84 or 168 mg for a person weighing 70 kg, tested on 92 or 93 study participants, NCT00143611). The daily total dose used in those trials exceeds the dose used here by nearly 500,000-fold. Results of the study have been published (CIT). The side effect of methemoglobinemia: "In the TAK-242 1.2 mg/kg/day group, mean levels increased from 0.9% at baseline to 2.8% at 2 hrs" appears to be of limited relevance for the 500,000-fold lower dose. Therefore, it is assumed that there will be no adverse effects. Biological activity of Resatorvid against LPS activity has been shown using human TLR4 and its co-receptors CD14 and MD2 expressed in HEK293 cells (CIT). The IC50 for LPS-induced NF-κB activation was found to be 110 nM. Assuming a dilution factor of about 10-fold upon intradermal injection and aiming for a receptor occupancy of at least 90%, using ~ 100-fold the IC50 was considered reasonable. Resatorvid (CAS 243984-11-4) is obtained from MedChemExpress, dissolved as 1 mM stock solution in DMSO and diluted to the final concentration of 10 µM, resulting in a solution containing 1% DMSO.

Azeliragon This RAGE antagonist is co-injected with LPS at a dose of 2 x 2.66 µg = 5.32 µg. Azeliragon has also undergone Phase III trials (daily dose of 5 mg orally for 18 months in ~440 study participants), where the daily total dose used exceeded the dose used here by nearly 1,000- fold (NCT02080364). It is also assumed here that there will be no adverse effects. Biological activity of 4 mg/kg intraperitoneal Azeliragon has been demonstrated by the reduction of LPS-induced airway inflammation (CIT). Binding of the prototypical RAGE agonist S100b is inhibited by Azeliragon with an IC50 of ~1 µM (International Publication Number WO2005000295). Assuming a dilution factor of about 10-fold upon intradermal injection and aiming for a receptor occupancy of at least 90%, using ~ 100-fold the IC50 was considered reasonable. Azeliragon (CAS 603148-36-3) is obtained from Targetmol, dissolved as 10 mM stock solution in DMSO and diluted to the final concentration of 100 µM, resulting in a solution containing 1% DMSO.

BCTC (N-(4-tert-butylphenyl)-4-(3-chloropyridin-2-yl)piperazine-1-carboxamide) This TRPV1 antagonist is administered at a total dose of 2 x 0.34 µg = 0.68 µg and added to the acidic solution. BCTC has been used in three previous studies at total doses of up to 3.36 µg per participant (CITs). No adverse effects were observed. The total dose of BCTC to be used here is approximately 20% of the previous maximal dose, so the risk of adverse effects is still considered very low. BCTC (CAS 393514-24-4) is obtained from Cayman Chemical and dissolved as 10 mM stock solution in DMSO. Solutions injected at timepoint 1 have a final DMSO concentration of 1%. Solutions containing final concentrations of Resatorvid, Azeliragon, BCTC and control were measured to have <0.01 Endotoxin Units/ml by a Limulustext according to the European Medicines Agency ICH Guideline Q4B. Passing through a 0.22 µm filter is used to obtain sterile solutions as a final step for all solutions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Full legal capacity

Exclusion Criteria:

* Participant of another study, ongoing or within the last four weeks
* Current medication intake (except hormonal contraception) or drug abuse
* Female subjects: Positive pregnancy test or breastfeeding
* Body temperature above 38°C, diagnostically verified
* Known allergic diseases, in particular asthmatic disorders and skin diseases
* Sensory deficit, skin disease or hematoma of unknown origin in the physical examination of the test site
* Symptoms indicating respiratory tract infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Skin Perfusion | 4.5h after the (non-)LPS injections
  The degree of hyperemia, quantified by laser speckle imaging, will be analyzed using ImageJ. The following steps describe the protocol for analyzing the (non-)inflamed spots of one forearm of a subject. To determine the volume under the surface (VUS, in analogy to an area under the curve, but for a 2-dimensional signal) of the flux change, for each of the previously injected skin spots a ROI covering the flow increase is adapted. The flux change (Δflux) is determined by subtracting from the average of the ROI the average signal of the surrounding forearm, and multiplying this with the ROI area. Any widespread or systemic change, which is not expected to occur, would be present in both the test site and the surrounding forearm and would therefore be corrected for by the chosen analysis approach. The analyzing person will be blinded concerning the type of injection. The variable is measured in arbitrary units (A.U.).

SECONDARY OUTCOMES:
Pain AUC | Between 4.5h and 5.5h after the (non-)LPS injections
  The outcome variable for (non-)acidic injections is based on pain ratings (0 = no pain, 100 = maximum imaginable pain), which are provided by the subjects every 5 seconds during and after the injections. Ratings continue until the participant reports zero pain for 30 consecutive seconds. The Area Under the Curve (AUC) of pain is calculated over the time span from 90 to 110 seconds (last 20 seconds or last 5 pain ratings of the acid injection). This yields the outcome variable 'Pain AUC'.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including pain ratings, time- stamped injection responses, and basic demographics (age, sex), will be shared after publication of the primary results. Only data used in the main publication and relevant supplementary analyses will be included.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be made available at the time of publication of the primary results article, as a supplementary file.
Access Criteria: All individuals who have access to the published article will be able to access the individual participant data (IPD) and supporting information as supplementary material. No special request or data use agreement is required.

REFERENCES:
- [Background] Schwarz MG, Namer B, Reeh PW, Fischer MJM. TRPA1 and TRPV1 Antagonists Do Not Inhibit Human Acidosis-Induced Pain. J Pain. 2017 May;18(5):526-534. doi: 10.1016/j.jpain.2016.12.011. Epub 2017 Jan 3. PMID 28062311
- [Background] Li J, Wang K, Huang B, Li R, Wang X, Zhang H, Tang H, Chen X. The receptor for advanced glycation end products mediates dysfunction of airway epithelial barrier in a lipopolysaccharides-induced murine acute lung injury model. Int Immunopharmacol. 2021 Apr;93:107419. doi: 10.1016/j.intimp.2021.107419. Epub 2021 Feb 3. PMID 33548580
- [Background] Kawamoto T, Ii M, Kitazaki T, Iizawa Y, Kimura H. TAK-242 selectively suppresses Toll-like receptor 4-signaling mediated by the intracellular domain. Eur J Pharmacol. 2008 Apr 14;584(1):40-8. doi: 10.1016/j.ejphar.2008.01.026. Epub 2008 Feb 5. PMID 18299127
- [Background] Rice TW, Wheeler AP, Bernard GR, Vincent JL, Angus DC, Aikawa N, Demeyer I, Sainati S, Amlot N, Cao C, Ii M, Matsuda H, Mouri K, Cohen J. A randomized, double-blind, placebo-controlled trial of TAK-242 for the treatment of severe sepsis. Crit Care Med. 2010 Aug;38(8):1685-94. doi: 10.1097/CCM.0b013e3181e7c5c9. PMID 20562702
- [Background] Kiers D, Leijte GP, Gerretsen J, Zwaag J, Kox M, Pickkers P. Comparison of different lots of endotoxin and evaluation of in vivo potency over time in the experimental human endotoxemia model. Innate Immun. 2019 Jan;25(1):34-45. doi: 10.1177/1753425918819754. PMID 30782041
- [Background] Suffredini AF, Hochstein HD, McMahon FG. Dose-related inflammatory effects of intravenous endotoxin in humans: evaluation of a new clinical lot of Escherichia coli O:113 endotoxin. J Infect Dis. 1999 May;179(5):1278-82. doi: 10.1086/314717. PMID 10191237
- [Background] Bretag AH. Synthetic interstitial fluid for isolated mammalian tissue. Life Sci. 1969 Mar 1;8(5):319-29. doi: 10.1016/0024-3205(69)90283-5. No abstract available. PMID 5781321
- [Background] Heber S, Ciotu CI, Hartner G, Gold-Binder M, Ninidze N, Gleiss A, Kress HG, Fischer MJM. TRPV1 antagonist BCTC inhibits pH 6.0-induced pain in human skin. Pain. 2020 Jul;161(7):1532-1541. doi: 10.1097/j.pain.0000000000001848. PMID 32107360
- [Background] Nair M, Jagadeeshan S, Katselis G, Luan X, Momeni Z, Henao-Romero N, Chumala P, Tam JS, Yamamoto Y, Ianowski JP, Campanucci VA. Lipopolysaccharides induce a RAGE-mediated sensitization of sensory neurons and fluid hypersecretion in the upper airways. Sci Rep. 2021 Apr 16;11(1):8336. doi: 10.1038/s41598-021-86069-6. PMID 33863932
- [Background] Yamamoto Y, Harashima A, Saito H, Tsuneyama K, Munesue S, Motoyoshi S, Han D, Watanabe T, Asano M, Takasawa S, Okamoto H, Shimura S, Karasawa T, Yonekura H, Yamamoto H. Septic shock is associated with receptor for advanced glycation end products ligation of LPS. J Immunol. 2011 Mar 1;186(5):3248-57. doi: 10.4049/jimmunol.1002253. Epub 2011 Jan 26. PMID 21270403
- [Background] Buters TP, Hameeteman PW, Jansen IME, van Hindevoort FC, Ten Voorde W, Grievink HW, Schoonakker M, de Kam ML, Gilroy DW, Feiss G, Rissmann R, Jansen MAA, Burggraaf J, Moerland M. Clinical, Cellular, and Molecular Effects of Corticosteroids on the Response to Intradermal Lipopolysaccharide Administration in Healthy Volunteers. Clin Pharmacol Ther. 2022 Apr;111(4):964-971. doi: 10.1002/cpt.2516. Epub 2022 Jan 6. PMID 34935141
- [Background] Buters TP, Hameeteman PW, Jansen IME, van Hindevoort FC, Ten Voorde W, Florencia E, Osse M, de Kam ML, Grievink HW, Schoonakker M, Patel AA, Yona S, Gilroy DW, Lubberts E, Damman J, Feiss G, Rissmann R, Jansen MAA, Burggraaf J, Moerland M. Intradermal lipopolysaccharide challenge as an acute in vivo inflammatory model in healthy volunteers. Br J Clin Pharmacol. 2022 Feb;88(2):680-690. doi: 10.1111/bcp.14999. Epub 2021 Aug 24. PMID 34293819